CLINICAL TRIAL: NCT04968522
Title: Attention Management Trial for Children With FASD - a N-of-1 Control Trial of Prescribed Stimulants for ADHD in FASD
Brief Title: FASST - Fetal Alcohol Spectrum Stimulant Trial
Acronym: FASST
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Monash Medical Centre (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, Alison Crichton, Principal Investigator, Monash Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RES-21-0000-248A; RES-21-0000-248A (Other: Monash Health HREC)
Record Dates: First submitted 2021-06-02; First posted 2021-07-20 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: Attention Deficit Hyperactivity Disorder; Stimulants; Trial; Attention
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders; Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Amphetamine

STUDY DESIGN:
Intervention Model Description: The N-of-1 trial has a four-period crossover design, comparing attention skills on active drug compared to placebo. The 8-week trial comprises four 2-week treatment blocks (each block consisting of 1 week active drug and 1 week placebo). Participants randomisation will be in the two-week pairs - so the order of treatment (A) and placebo (P) to be randomly assigned within each two-week cycle is randomly allocated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The order of medications (placebo/active drug) will be masked to the participant, assessors and investigator. At the end of the trial, the order of medications will be unmasked, and compared with the parent and teachers' observations of the child's behaviour.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo comparator 2 (Placebo Comparator): Participants will be allocated a randomly allocated sequence of treatment. The randomisation will be in two-week pairs - so the order of treatment (A) and placebo (P) to be randomly assigned within each two-week cycle (over 8 weeks). Placebo will be matched in dose to their stimulant dose at enrolment to the trial as determined and titrated by their primary paediatrician. This dose will remain constant for the course of the trial (8 weeks). Placebo will be orally administered, unless this is not possible for clinical reasons.
  Interventions: Drug: Placebo
- Stimulant (Experimental): The stimulants used in the trial are commercially available and will be used in accordance with the approved labelling. Participants must be on a stable dose of stimulant medication for at last 1 month prior to the study. The dose is individualized and titrated by treating primary paediatrician. This will represent the starting dose for the trial, and this will remain stable through the course of the 8-week trial. This study is a N-of-1 RCT of currently prescribed stimulant medications for treatment of ADHD symptoms in children with FASD, relative to matched placebo capsules. Based on pilot data from this group, psychostimulant medications prescribed in this population may include:
  * Methylphenidate IR
  * Methylphenidate LA
  * Dexamphetamine
  Children will take the required number of capsules to match the total prescribed dose (e.g. 30mg Ritalin LA is 3x10mg capsules).
  Interventions: Drug: Methylphenidate Hydrochloride; Drug: Methylphenidate Hydrochloride 18 MG; Drug: Dexamphetamine sulfate

INTERVENTIONS:
Drug: Methylphenidate Hydrochloride — This study is a N-of-1 RCT of currently prescribed stimulant medications for treatment of ADHD symptoms in children with FASD, relative to matched placebo capsules. The Ritalin 10 will be administered at the child's prescribed dose and may include a half tablet (5mg) increment. Ritalin 10 will be encapsulated in full tablet (10mg) or half tablet (5mg) dose.
  Other Names: Ritalin 10 tablets
  Arms: Stimulant
Drug: Placebo — The placebo is Maize Starch and Pregelatinised Maize Starch. The placebo will be encapsulated using the same capsule that is opaque so that participants cannot distinguish the two visually. Where the active mediation amount is small for the capsule, there will be additional Starcke 1500 (Maize Starch and Pregelatinised Maize Starch) added to fill the capsule so that the active drug and capsule also weigh approximately the same. The dose of placebo will be matched to the participants currently prescribed stimulant medication.
  Arms: Placebo comparator 2
Drug: Methylphenidate hydrochloride — This study is a N-of-1 RCT of currently prescribed stimulant medications for treatment of ADHD symptoms in children with FASD, relative to matched placebo capsules. The Ritalin LA will be administered at the child's prescribed total dose. Ritalin LA will be encapsulated.
  Other Names: Ritalin LA Long acting capsules
  Arms: Stimulant
Drug: Methylphenidate Hydrochloride 18 MG — This study is a N-of-1 RCT of currently prescribed stimulant medications for treatment of ADHD symptoms in children with FASD, relative to matched placebo capsules. The Concerta (18mg) will be administered at the child's prescribed total dose. Concerta will be encapsulated.
  Other Names: Concerta
  Arms: Stimulant
Drug: Dexamphetamine sulfate — This study is a N-of-1 RCT of currently prescribed stimulant medications for treatment of ADHD symptoms in children with FASD, relative to matched placebo capsules. The Dexamphetamine (10mg) will be administered at the child's prescribed total dose. Dexamphetamine will be encapsulated.
  Other Names: Aspen Dexamfetamine Tablets
  Arms: Stimulant

SUMMARY:
This study is a double-blind, placebo controlled, series of N-of-1 trials of individualised stimulant dose on ADHD symptomatology in children with FASD.

The broad aim of this study is to contribute new evidence towards understanding treatment efficacy for ADHD symptoms in FASD.

Specific aims are:

1. To assess the ongoing effectiveness of stimulant medication prescribed for ADHD symptoms in individual children with FASD of clinically prescribed stimulant medication compared to placebo to control ADHD symptoms (using behavioural and cognitive measures) in children with FASD and ADHD using a N-of-1 trial design.
2. To obtain pilot data to examine feasibility and tolerability of the planned N-of-1 trial design in children with FASD and ADHD for future and larger studies that might seek to examine if the different stimulant types are equally effective relative to placebo.
3. To review the multiple N-of-1 data to analyze key individual factors that mediate the effect of stimulants relative to placebo on ADHD symptoms, including underlying child factors (attention skills, cognitive function), sociodemographic factors and other prenatal exposures.

DETAILED DESCRIPTION:
Study Design:

This is a single site, double-blind, placebo controlled, N-of-1 trial of clinically prescribed, individualised stimulant dose on ADHD symptomatology in children with FASD. The N-of-1 trial has four 2-week treatment blocks (each block consisting of 1 week active drug and 1 week placebo). Interventions will include either prescribed stimulant (active drug) or matched placebo capsules, compared in four 2-week treatment blocks (each block consisting of 1 week active drug and 1 week placebo). Participants will be randomized to the sequence of the treatment arms. Randomisation will be in the two-week pairs - so the order of treatment (A) and placebo (P) to be randomly assigned within each two-week cycle.

Secondarily the investigators will collate outcomes across the N-of-1 trials and make use of a 'series' or multiple N-of-1 trial design18, chosen as it is a valid method of trial design for rare clinical disorders where individualized treatments are required. This design can result in robust evidence, assuming standards of methodological practice.1 In an N-of-1 trial, each participant is assured of receiving both the study medication and placebo, and thus learns whether the treatment works specifically for them or not.

Study objectives:

1. Primary objective:

   Test ongoing effectiveness of stimulant medication in individual children with FASD on pharmacotherapy for ADHD symptomatology, using individual N-of-1 trials.
2. Secondary objectives:

Secondary objective 1: To examine feasibility and tolerability of the N-of-1 trial design in children with FASD and ADHD for future, larger studies that might seek to examine if the different stimulant types are equally effective relative to placebo.

Secondary objective 2: Through quantitative analysis of a series of N-of-1 trials,1 explore individual factors that mediate the effect of stimulants relative to placebo on ADHD symptoms, on children with FASD, including underlying attention skills, cognitive function and other child/sociodemographic factors and additional prenatal exposures.

Exploratory objectives: Investigators will review if there is any change in pediatrician patient management post trial.

Study Population:

Children (4-18 years) with FASD and ADHD seen by the Victorian Fetal Alcohol Service (VicFAS), prescribed stimulant medication for ADHD symptoms. The age limit selected was based on the age in which stimulants have been shown to be effective in controlling ADHD symptoms in the general population, and who are seen by the clinical service.

VicFAS assesses 20 children per year at the diagnostic clinic. All participants are currently approached for consent to the already established VicFAS database, which includes full child demographic, clinical and neurodevelopmental information as well as optional consent for future studies. Participants who have consented to this optional inclusion will be re-consented to this study.

A total of 20 participants will be approached for recruitment to the study. This will be a convenience sample of children seen through the VicFAS FASD diagnostic clinic since inception in September 2019 until study completion (n=20).

Each participant will undergo repeated measures. Estimation of the needed number of cross-overs (that is 'sample size' in N-of-1 studies) was based on having at least 80% power (β = 0.20) to detect a 5.9-point reduction. With 36 observations per participant, (18 placebo, 18 active medication) we achieve >80% power (alpha of 0.05 will be used as the cut-off for significance, one-sided hypothesis test).

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be enrolled in this trial:

* Is between the ages of 4 - 18 years at the time of randomization.
* Meet diagnostic criteria for FASD or at risk of FASD according to the Australian Guide to the diagnosis of FASD.
* Is a patient of VicFAS or Developmental Paediatrics (Monash Health).
* Has a diagnosis of ADHD according to the DMS-IV criteria.
* Be on a stimulant medication for treatment of ADHD symptoms.
* Be on a stimulant medication as a primary treatment for ADHD.
* Be on a stable dose of stimulant medication for at last 1 month prior to the study.
* Provide a signed and dated informed consent form / and has a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf.
* If seen by VicFAS/Developmental paediatrics between August 2019 - study commencement date), parent/guardian must have provided verbal or written consent to the VicFAS database PICF and selected 'yes' to the optional consent for contact for 'future research'.

Exclusion Criteria:

Exclusion criteria will include any of the following:

* Inability to read or speak sufficient English for either child or parent/guardian to complete assessment tasks.
* Be on a medication for treatment of ADHD symptoms that is a medication other than stimulants as a primary treatment for ADHD.
* Allergy/sensitivity to Starcke 1500 (Maize Starch and Pregelatinised Maize Starch).
* Unable to swallow capsules.
* Intracranial symptoms or pathology such as epilepsy, hydrocephalus, diagnosed traumatic. brain injury or progressive intracranial tumours that may impact cognitive and behavioural function (children with asymptomatic or static lesions will be eligible).
* An abnormal ECG result at the time of screening deemed clinically significant by study physician.
* Presence of a significant comorbid psychiatric or psychological (excluding ADHD, oppositional defiant disorder, conduct disorder and pervasive development disorder/autism spectrum disorder) including depressive disorder, anxiety disorder, psychotic disorder, suicidality, Tic disorder, anorexia or bulimia nervosa
* Has a known hypersensitivity to starch or other compound relevant to placebo/capsules.
* Has had treatment with any other investigational drug within 4 weeks prior to randomisation.
* If the participant is known to be pregnant, they cannot take part in this research project.
* Parent/guardian not consenting to contact with paediatrician or school.
* Is deemed by their treating paediatrician to be medically unsafe for trial participation.
* Child's school unwilling to participate in outcome assessments.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD symptoms - teacher report - between placebo and stimulant | Daily for 5 week days (Monday - Friday) of each trial week (8 weeks total)
  ADHD symptoms will be measured using the Conners 3rd Edition-Teacher (Conners 3-T), for 6-18 year old's and the Conners Early Childhood teachers/childcare providers (full length) form for participants 2-6 years. Each item is rated on a Likert scale from 0 to 3 (0=never or rarely; 1=sometimes; 2=often; 3=very often). Test- retest values for the Conners scales indicate excellent temporal stability (ranging from .73 to 1.00).
  The T-score is norm referenced, with a mean of 50. The average range falls within one standard deviation of the mean (i.e., between 40 and 59). A higher score indicates more elevated symptoms. T score Guideline 70+Very Elevated Score 65-69 Elevated Score 40-59 Average score 60-64 High average score < 40 Low score. Investigators will examine Inattentive and Hyperactivity/Impulsivity Symptom Scales. Symptoms indicated for each subscale are summed to get total.
Change in ADHD symptoms - parent report - between placebo and stimulant | Daily for 5 week days (Monday - Friday) of each trial week (8 weeks total)
  ADHD symptoms will be measured using the Conners 3rd Edition-Parent (Conners 3-P), for 6-18 year old's and the Conners Early Childhood parent (full length) form for participants 2-6 years. Each item is rated on a Likert scale from 0 to 3 (0=never or rarely; 1=sometimes; 2=often; 3=very often). Test- retest values for the Conners scales indicate excellent temporal stability (ranging from .73 to 1.00).
  The T-score is norm referenced. The average range falls within one standard deviation of the mean (i.e., between 40 and 59). A higher score indicates more elevated symptoms. T score Guideline 70+Very Elevated Score 65-69 Elevated Score 40-59 Average score 60-64 High average score < 40 Low score. Investigators will examine Inattentive and Hyperactivity/Impulsivity Symptom Scales. Symptoms indicated for each subscale are summed to get the total.
Change in spatial working memory - between placebo and stimulant | Day 3 of each trial week (8 weeks total)
  Spatial Working Memory (SWM) task from the Cambridge Neuropsychological Test Automated Battery. SWM is a component of cognitive executive function which is measured by SWM task of CANTAB between the errors. The ability to retain spatial information and manipulate remembered items in working memory will be measured with the SWM task of CANTAB which is self-ordered and assesses the individual's ability to strategise. Between search errors will be analysed. Scores are raw scores, with no normative data available. Higher error score indicated poorer performance. Scale does not have a maximum range.
Change in Visual Information Processing - between placebo and stimulant | Day 3 of each trial week (8 weeks total)
  Rapid Visual Information Processing (SOC) from Cantab. SOC Stockings of Cambridge (SOC) is a test of spatial planning that requires individuals to use problem-solving strategies to match two sets of stimuli. The participant must move the balls in the bottom display to copy the pattern shown in the top display. The balls are moved one at a time by selecting the required ball, then selecting the position to which it should be moved. The participant is instructed to make as few moves as possible to match the two pattern.
  The outcome measure of this subtest is the number of problems completed, regardless of whether the maximum moves limit was reached on any problem.

SECONDARY OUTCOMES:
Change in child problem behaviour rating- between placebo and stimulant | Daily for 5 week days (Monday - Friday) of each trial week (8 weeks total)
  Top Problem Rating. This will be used as a brief but robust measure of child emotional and behavioural difficulties as rated by the parent. Top Problems Assessment (TPA) is a brief, idiographic procedure that allows clinicians and researchers to identify problems of children that are especially important from the perspective of the caregiver. The severity of these problems, once identified, will monitored daily.
  The overall severity of problem rating (0 - 4) between placebo and active medication arms will be used as an indicator of problem worsening or improving. as one index of whether improvement is occurring. A higher problem rating indicates greater perceived difficulties.
Change in functional Impairment- between placebo and stimulant | Daily for 5 week days (Monday - Friday) of each trial week (8 weeks total)
  Impairment resulting from ADHD symptoms. This scale contains the items that are most likely to represent the participant's target of treatment. The instrument uses a Likert scale such that any item rating 2 or 3 is clinically impaired. The scale is scored generating the total score. When defining impairment for DSM-IV, any domain with at least two items scored 2, one item scored 3 or a mean score >1.5 is impaired.
Difference in side effects during placebo and stimulant phase | Day 5 of each trial week (8 weeks total)
  Investigators will monitor side effects of the placebo and active medication using the Barkley Side Effects Rating Scale (17 symptoms; 0 = absent, severity rated from 1 to 9). Parent ratings of side effects for the drug and placebo conditions will be described using the mean total side effect rating for each condition.
Trial feasibility - recruitment rate | End of 8 month active trial phase
  Feasibility of the study (n-of-1 design) will be explored using trial recruitment rate across the trial from study start to study close. Investigators will calculate recruitment feasibility as the percentage of eligible participants agreeing to participate. A higher percentage will indicate greater participation.
Trial feasibility - completion rate | End of 8 month active trial phase
  Feasibility of the study (n-of-1 design) will be explored using completion rates across the trial from study start to study close. Completion rate will be the percentage of enrolled participants who complete the trial. A higher percentage will indicate greater participation.
Compliance | End of 8 month active trial phase
  Investigators will inspect participant medication diaries, to calculate treatment compliance. Non-compliance will be defined as missing more than one or more days of the active drug or placebo condition.
Assessment completion rate | End of 8 month active trial phase
  Investigators will calculate the percentage of outcome assessments completed by each participant to examine assessment feasibility of the study design.
Data completion reason | End of 8 month active trial phase
  Investigators will also examine reasons for incomplete outcome data.
Adverse events | End of 8 month active trial phase
  Adverse events (AE's) will be coded using the, Medical Dictionary for Regulatory Activities (MedDRA), and calculated once each per participant. We will describe the total number of AE's across the trial.

OTHER OUTCOMES:
Rate of change of prescribed stimulant | End of trial (8 weeks)
  Participant's paediatrician will rate any change in medication practice, immediately post-trial. This will capture the rate of this change in medication as a result of the N-of-1 trial data over the whole study.
Attention Deficit Hyperactivity Disorder subtype classification | Baseline
  Conners 3 parent and teacher ratings will be used to classify child ADHD subtype (ADHD inattentive type, ADHD Hyperactive-Impulsive type, ADHD Combined type) according to DMS related symptom count cut-offs (At least 6 out of 9 symptoms) for each subtype or combined type.
Attention factor 1 (selective) | Baseline
  The Tea-Ch measures four factors of child attention. Selective, or focused attention will be measures using the Sky Search task. This measure provides both raw score and scaled scores for each of the subtests. We will use age and gender based scaled scores for selective attention outcome. Scaled scores have a mean of 10 and standard deviation of 2. A lower score indicates greater impairment in the attentional factor.
Attention factor 2 (sustained) | Baseline
  The Tea-Ch measures four factors of child attention. Sustained attention will be measures using the Score! task. This measure provides both raw score and scaled scores for each of the subtests. We will use age and gender based scaled scores for sustained attention outcome. Scaled scores have a mean of 10 and standard deviation of 2. A lower score indicates greater impairment in the attentional factor.
Attention factor 3 (divided) | Baseline
  The Tea-Ch measures four factors of child attention. Switching attention will be measures using the Sky Search DT task. This measure provides both raw score and scaled scores for each of the subtests. We will use age and gender based scaled scores for divided attention outcome. Scaled scores have a mean of 10 and standard deviation of 2. A lower score indicates greater impairment in the attentional factor.
Attention factor 4 (alternating) | Baseline
  The Tea-Ch measures four factors of child attention. Alternating attention (i.e. switching focus from one stimuli to another) will be measures using the Creature counting task. This measure provides both raw score and scaled scores for each of the subtests. We will use age and gender based scaled scores for alternating attention outcome. Scaled scores have a mean of 10 and standard deviation of 2. A lower score indicates greater impairment in the attentional factor.
Cognitive ability level | Baseline
  Child intellectual functioning will be assessed at baseline using age based normed Full Scale IQ from age appropriate Weschler scales (WPPSI-IV or WISC-V). The median Full Scale IQ is centered at 100, with a standard deviation of 15. A higher score indicates greater cognitive ability.
Domains of neurodevelopmental impairment | Baseline
  Children's overall level of neurodevelopmental impairment will be calculated by tallying the total number of domains assessed as significantly impaired (<3rd percentile on a standardised measures) against Australian FASD diagnostic criteria (0-10), including: Brain structure and neurology, motor skills, cognition, language, academic achievement, memory, attention, executive function, affect regulation and adaptive behaviour/social communication. The total number of domains impaired is added up for each participant using domain specific criteria (See FASD guide), defined by performance below the third percentile. The range is 0-10; a higher count is greater number of domains of impairment.
Demographics | Baseline
  Child demographic (age, sex) data will be extracted from medical records.
Socioeconomic status | Baseline
  Family details and socioeconomic status will be coded from medical record review: ethnic group mother & child, child language spoken at home, parental relationship status, family structure (custody), number of children living in household, maternal work status, socioeconomic status (postcode).

CONTACTS AND LOCATIONS:
Overall Officials: Alison Crichton, PhD, Principal Investigator — Monash Children's Hospital
Locations (1):
- Monash Health, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Beginning 3 months following analysis and article publication, the following will be made available long-term for use by future researchers from a recognised research institution whose proposed use of the data has been ethically reviewed and approved by an independent committee and who accept Monash Health institutional conditions for access:
  * Group level data that underlie the results reported in this article after de-identification (text, tables, figures and appendices)
  * Trial protocol, PICF

REFERENCES:
- [Derived] Crichton A, Harris K, McGree JM, Nikles J, Anderson PJ, Williams K. Fetal alcohol spectrum disorder and attention deficit hyperactivity disorder stimulant trial in children: an N-of-1 pilot trial to compare stimulant to placebo (FASST): protocol. BMJ Open. 2024 Apr 17;14(4):e071266. doi: 10.1136/bmjopen-2022-071266. PMID 38631835